CLINICAL TRIAL: NCT06485557
Title: A Prospective Cohort Study of Neoadjuvant Chemotherapy Plus Sintillumab in the Treatment of Resectable NSCLC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIT20240507
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Resectable Non-small Cell Lung Cancer
Keywords: NSCLC; Neoadjuvant; Sintillumab
MeSH Terms: interventions — sintilimab; Platinum Compounds

STUDY DESIGN:
Intervention Model Description: A Prospective Cohort Study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A (Experimental): receive 3 cycles of sintilimab plus platinum-based chemotherapy
  Interventions: Drug: sintilimab plus platinum-based chemotherapy
- group B (Experimental): receive 2 cycles of sintilimab plus platinum-based chemotherapy plus 1 cycle of sintilimab
  Interventions: Drug: sintilimab plus platinum-based chemotherapy
- group C (Experimental): receive 1 cycle of sintilimab plus platinum-based chemotherapy plus 2 cycles of sintilimab
  Interventions: Drug: sintilimab plus platinum-based chemotherapy

INTERVENTIONS:
Drug: sintilimab plus platinum-based chemotherapy — The subjects in group A will receive 3 cycles of sintilimab plus platinum-based chemotherapy
  Other Names: Group A
  Arms: group A
Drug: sintilimab plus platinum-based chemotherapy — The subjects in group B will receive 2 cycles of sintilimab plus platinum-based chemotherapy plus 1 cycle of sintilimab
  Other Names: Group B
  Arms: group B
Drug: sintilimab plus platinum-based chemotherapy — The subjects in group C will receive 1 cycle of sintilimab plus platinum-based chemotherapy plus 2 cycles of sintilimab.
  Other Names: Group C
  Arms: group C

SUMMARY:
This study uses a prospective cohort design.Subjects are randomly divided into three groups (A, B, C) before surgery. Group A gets 3 cycles of sintilimab + chemo, Group B gets 2 cycles + 1 cycle, and Group C gets 1 cycle + 2 cycles.

Non-squamous NSCLC subjects receive pemetrexed/albumin paclitaxel + platinum, while squamous NSCLC subjects get albumin paclitaxel + platinum.

DETAILED DESCRIPTION:
This study adopts a prospective cohort study design.The subjects will be randomly divided into three groups according to the ratio of 1:1:1 prior to surgery: group A, group B and group C. The subjects in group A will receive 3 cycles of sintilimab plus platinum-based chemotherapy, group B will receive 2 cycles of sintilimab plus platinum-based chemotherapy plus 1 cycle of sintilimab, and group C will receive 1 cycle of sintilimab plus platinum-based chemotherapy plus 2 cycles of sintilimab. Non-squamous NSCLC subjects will receive pemetrexed/albumin paclitaxel and platinum (cisplatin/carboplatin), and squamous NSCLC subjects will receive albumin paclitaxel and platinum (cisplatin / carboplatin).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign the written informed consent form (ICF), and be able to follow the visits and relevant procedures specified in the protocol
2. Age ≥ 18 years
3. Cytologically or histologically confirmed primary NSCLC (including adenocarcinoma, squamous cell carcinoma, adenosquamous carcinoma)
4. Subjects with Stage IIA (primary focus>4cm), IIIA or IIIB (resectable N2 only) disease based on the 8th edition of the TNM staging classification for lung cancer issued by the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification (AJCC8), resectable N2 only refers to non-massive (defined as short diameter less than 3cm), discrete or single station N2 involvement.
5. No EGFR sensitive mutations and ALK rearrangements should be tested in non-squamous non-small cell lung cancer, and will be not mandatory in squamous cell carcinoma
6. Deemed radically resectable with curative intent
7. Pulmonary function reached the standard of planned pneumonectomy ( FEV1 ≥ 50 % predicted value, MVV ≥ 50 % predicted value ), and there was no surgical contraindication
8. Enough tissue samples for PD-L1 detection (Number of slices ≥ 6)
9. At least one measurable lesion in line with RECIST V1.1
10. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
11. Have not received any prior systemic anti-tumor therapy or local radiotherapy for NSCLC
12. Have adequate organ and bone marrow function, and the laboratory examination values within 14 days prior to enrollment meet the following requirements (no blood components, cell growth factors, albumin and other intravenous or subcutaneously administered drugs to correct hematological or liver and kidney dysfunction were allowed within the first 14 days of obtaining laboratory tests), as follows:
13. Hematological function was sufficient, defined as absolute neutrophil count ≥ 1.5 × 109 / L, platelet count ≥ 100 × 109 / L, hemoglobin ≥ 100g / L;
14. Full liver function, defined as total bilirubin level ≤ 1.5 × ULN, AST and ALT level ≤ 2.5 × ULN, albumin (ALB) ≥ 35g / L;
15. Renal function was sufficient, serum creatinine (Scr) ≤ 1.5 × ULN, creatinine clearance rate (CrCl) ≥ 60mL / min (calculated by Cockcroft / Gault formula) and urine routine test results showed that urinary protein (UPRO) < 2 + or 24-hour urinary protein < 1g;
16. The international normalized ratio (INR) ≤ 1.5 × ULN, and prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN within 7 days before treatment;
17. For women of childbearing age, urine or serum pregnancy tests were negative for at least seven days prior to the first study drug administration. If the urine pregnancy test is positive, a blood pregnancy test is required;
18. If there is a risk of conception, male and female patients need to use high-efficiency contraception (i.e., the method with an annual failure rate of less than 1 %) and continue until at least 180 days after discontinuation of the trial; Note: If abstinence is the normal lifestyle and preferred contraceptive method of the subjects, abstinence can be accepted as a contraceptive method.

Exclusion Criteria:

1. Pathological examination showed that small cell carcinoma, neuroendocrine carcinoma, sarcoma, lymphoepithelioma-like carcinoma, salivary gland tumor and mesenchymal tumor components
2. Tumor invasion of the diaphragm, mediastinum, heart, pericardium, large blood vessels (such as aorta), esophagus, vertebral body
3. pulmonary sulcus tumor
4. Contralateral lung nodules, it need biopsy if clinically suspected
5. Subjects with confirmed or suspected brain metastases
6. Currently participating in an interventional clinical study or treatment with another study drug or study device within 4 weeks prior to randomization
7. Previous use of anti-PD-1, anti-PD-L1, anti-programmed death receptor ligand 2 (PD-L2) or anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) drugs or any other drugs acting on T cell co-stimulation or immune checkpoint pathways (such as OX40, CD137, etc.) and adoptive cellular immunotherapy
8. Received drugs with immunomodulatory effects (including thymosin, interferon, interleukin) within the first 4 weeks of randomization
9. Received live attenuated vaccine within the first 4 weeks of randomization（Or plan to receive live attenuated vaccine during the study period） Note: Acceptance of inactivated vaccine for seasonal influenza is permitted; however, live attenuated influenza vaccine is not allowed
10. Need long-term systemic use of corticosteroids，received any other form of immunosuppressive therapy within 7 days before randomization Note: Nasal spray, inhalation or other local glucocorticoids or physiological doses of systemic glucocorticoids (≤ 10mg / day prednisone or equal doses of drugs) or for pretreatment (such as prevention of contrast agent allergy) use is allowed
11. A history of non-infectious pneumonia requiring glucocorticoid therapy or current interstitial lung disease (≥ grade 2) within the previous year of randomization
12. Active autoimmune diseases, including but not limited to inflammatory bowel disease, such as ulcerative colitis or Crohn 's disease, that require systemic treatment ( such as the use of disease-modifying drugs, corticosteroids or immunosuppressants ), have occurred within the first two years of the randomization; diverticulitis; chylous diarrhea; systemic lupus erythematosus; sarcoidosis syndrome or wegener syndrome ( granuloma with polyangiitis); graves' disease; rheumatoid arthritis; multiple sclerosis; vasculitis; glomerular nephritis; antiphospholipid syndrome; pituitary inflammation; uveitis, etc. Alternative therapies (such as thyroxine, insulin, or physiological doses of corticosteroids for adrenal or pituitary dysfunction) are not considered as systemic treatments. Patients with positive autoimmune antibodies need to be evaluated by researchers to confirm that there is no autoimmune disease that requires systemic treatment before they can be enrolled
13. Primary immunodeficiency disease
14. Previous or current myocarditis
15. Not fully recovered from toxicity and/or complications caused by any intervention before randomization (> grade 1 or not recovery to baseline)
16. peripheral neuropathy ≥ grade 2
17. Hereditary bleeding tendency or coagulation dysfunction, or a history of thrombosis: There have been any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism.within the previous 6 months of randomization. Have a history of deep vein thrombosis or any other serious thromboembolism (implantable venous access port or catheter-derived thrombosis, or superficial venous thrombosis is not considered thromboembolism) within the previous 3 months of randomization
18. Non-squamous NSCLC subjects who were unable or unwilling to receive folic acid or vitamin B12 supplementation
19. Any unstable systemic disease or concurrent disease, including but not limited to:

1）Active infection ( requiring anti-infective drugs or systemic anti-infective drugs used within the previous week of randomization ) ; 2）congestive heart failure [New York Heart Association, NYHA ≥ grade II]； 3）Severe arrhythmia, liver, kidney, or metabolic disease requiring medical treatment； 4）Untreated coronary atherosclerotic heart disease； 5）Have a history of gastrointestinal perforation and / or fistula, a history of intestinal obstruction, extensive bowel resection or long-term chronic diarrhea within the previous 6 months.

20.Received solid organ or blood system transplantation

21.Have a history of HIV infection (HIV1/2 antibody positive), active syphilis

22.Tuberculosis, which is active or requires medical intervention at this stage, including but not limited to pulmonary tuberculosis

23.Active Hepatitis B Subjects with hepatitis B who met the following criteria met the inclusion criteria: HBsAg (+) or HBcAb (+), HBV viral load < 2000 copies/ml or < 200 IU/ml or lower than the detection limit HBsAg Subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-) do not need to receive prophylactic anti-HBV treatment, but need to closely monitor whether the virus is reactivated

24.Active hepatitis C (HCV antibody positive and HCV-RNA level above the detection limit)

25.Patients with malignant tumors other than confirmed NSCLC within the first 5 years of randomization, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, and thyroid papillary carcinoma after radical surgery

26.Sintilimab and/or selected chemotherapy regimens (non-squamous NSCLC : pemetrexed plus cisplatin or carboplatin ; squamous NSCLC : Albumin paclitaxel plus cisplatin or carboplatin) active ingredients and/or any excipients have allergic reactions

27.Pregnant or lactating women or women preparing to be pregnant or lactating during the study period

28.Subjects are mental illness or drug abuse that may have an impact on compliance with the test requirements, and have a history of alcohol abuse

29.Subjects with medical history, disease, treatment or laboratory abnormality which may interfere with the results of the trial, prevent the subject from participating in the study throughout the study, or the researchers believe that subjects in the study can not get the best interests of the subject Local or systemic diseases caused by non-malignant tumors, or secondary reactions to cancer, can lead to higher medical risks and/or uncertainty in survival evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 4 months
  rate of pathological complete response

SECONDARY OUTCOMES:
MPR rate | 4 months
  rate of major pathologic response
R0 resectability rate | 4 months
  R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed
The completion rate of surgery on schedule | 4 months
  The rate of surgical completion as per the pre-established schedule represents a crucial metric in evaluating the efficiency and precision of medical institutions

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy